CLINICAL TRIAL: NCT03235128
Title: Clinical Significance of Assesment of Serum miRNA-30a in Childhood Nephrotic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAMahmoud, Principle investigator, Assiut University
Other Study IDs: CSOAOSM
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Nephrotic Syndrome Steroid-Resistant
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group1: Steroid sensitive nephrotic syndrome(10 cases).
  Interventions: Diagnostic Test: ‗Urine analysis ‗Urine protein quantification ‗Serum albumin ‗Lipid profile.Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood.
- Group2: Steroid resistant nephrotic syndrome(10 cases).
  Interventions: Diagnostic Test: ‗Urine analysis ‗Urine protein quantification ‗Serum albumin ‗Lipid profile.Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood.
- Group3: immunosuppressive resistant nephrotic syndrome(10 cases).
  Interventions: Diagnostic Test: ‗Urine analysis ‗Urine protein quantification ‗Serum albumin ‗Lipid profile.Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood.
- Group4: Refractory nephrotic syndrome(10 cases).
  Interventions: Diagnostic Test: ‗Urine analysis ‗Urine protein quantification ‗Serum albumin ‗Lipid profile.Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood.
- Group5: Normal children as a healthy control group(5 cases).
  Interventions: Diagnostic Test: ‗Urine analysis ‗Urine protein quantification ‗Serum albumin ‗Lipid profile.Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood.

INTERVENTIONS:
Diagnostic Test: ‗Urine analysis ‗Urine protein quantification ‗Serum albumin ‗Lipid profile.Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood. — Specific tests Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood

SUMMARY:
Childhood nephrotic syndrome is the most frequent glomerular disease that presents during childhood,primarily owing to a disturbed immune function.This disease is characterized by alterations in selectivity at the glomerular capillary wall that lead to an inability to restrict the urinary loss of protein.

DETAILED DESCRIPTION:
Childhood nephrotic syndrome is the most frequent glomerular disease that presents during childhood,primarily owing to a disturbed immune function.This disease is characterized by alterations in selectivity at the glomerular capillary wall that lead to an inability to restrict the urinary loss of protein.The syndrome is characterized by the tetrad of nephrotic range proteinuria (>40 mg/m2/hour), hypoalbuminemia (<2.5 g/dl), generalized edema, and hyperlipidemia. It can be congenital or acquired.Currently,serum albumin, lipids, and proteinuria are the common diagnostic markers of childhood NS, but these markers may not accurately predict the outcome of individual patients because of the heterogeneity of the disease. Renal biopsy is more precise for establishing prognosis of renal outcome, but it has potential complications. Repeated monitoring is technically difficult, particularly for children. Therefore, there is still an urgent need to identify new non invasive diagnostic and prognostic biomarkers and new therapeutic targets for this disease.miRNA-30a expression in the serum of patients with nephrotic syndrome and analyzed the correlation between miRNA with largest over expression level and clinical features compared with healthy subjects.miRNA-30a expression level in drug resistant nephrotic syndrome patients was obviously higher than the drug sensitive patients and up-regulated most significantly in mesangial proliferative glomerulonephritis among different pathological types, while it decreased most obviously in glomerular lesions. miRNA-30a could be treated as the molecular marker in predict drug resistance, pathological type of nephrotic syndrome and follow up of resistant cases.

ELIGIBILITY:
Inclusion Criteria:

-Nephrotic children aged from 2 to 18 that admitted to Pediatric Hospital.

Exclusion Criteria:

* Congenital or infantile nephrotic syndrome
* Other kidney diseases
* Abnormal kidney function test

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group1: steroid sensitive nephrotic syndrome ( 10 cases ). Group2:steroid resistant nephrotic syndrome (10 cases). Group3:immunosuppresive resistant nephrotic syndrome(10 cases). Group4:refractory nephrotic syndrome(10 cases). Group5: normal children as a healthy control group ( 5 cases ).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with highly expressed serum miRNA30-a in resistant cases of childhood nephrotic syndrome. | 3 days
  Quantitation of miRNA -30a by Real-time polymerase chain reaction (Q-PCR) in peripheral blood.

REFERENCES:
- [Background] Teng J, Sun F, Yu PF, Li JX, Yuan D, Chang J, Lin SH. Differential microRNA expression in the serum of patients with nephrotic syndrome and clinical correlation analysis. Int J Clin Exp Pathol. 2015 Jun 1;8(6):7282-6. eCollection 2015. PMID 26261628